CLINICAL TRIAL: NCT02726971
Title: A Prospective, Randomized, Controlled Trial Comparing 2 Different Doses of Estrogen Therapy After Hysteroscopic Adhesiolysis as an Adjuvant to Prevent Recurrence of Intrauterine Adhesions
Brief Title: Comparison of Different Doses of Oestrogen Therapy for Preventing Intrauterine Adhesion
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fu Xing Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Jun Guo, Chief Physician, Fu Xing Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LYuhuan
Record Dates: First submitted 2016-03-22; First posted 2016-04-04 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Asherman Syndrome
Keywords: Intrauterine Adhesion; Oestrogen Artificial Periodic Therapy
MeSH Terms: conditions — Gynatresia | interventions — femoston

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose of oestrogen (Experimental): Patients in this group will build artificial cycle by Femoston.(oral one red tablet daily for 11 days and oral one yellow tablet in the next 10 days). This process will last for 3 months after the surgery.
  P.S.1.A red tablet contains 2mg estradiol. 2.A yellow tablet contains 2mg estradiol and 10mg dydrogesterone.
  Interventions: Drug: Femoston
- High dose of oestrogen (Active Comparator): Patients in this group will build artificial cycle by Femoston.(oral three red tablets daily for 11 days and oral two yellow tablets in the next 10 days). This process will last for 3 months after the surgery.
  P.S.1.A red tablet contains 2mg estradiol. 2.A yellow tablet contains 2mg estradiol and 10mg dydrogesterone.
  Interventions: Drug: Femoston

INTERVENTIONS:
Drug: Femoston — Femoston is a Complex Packing Estradiol Tablets and Estradiol and Dydrogesterone.

SUMMARY:
This single-center,prospective,randomized,controlled trial is conducted to evaluate the efficacy of different doses of estrogen artificial periodic therapy after hysteroscopic adhesiolysis in patients with moderate-severe adhesion.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate and severe IUA according to the AFS IU adhesion scoring system (AFS 1988 version) (19) showed in Table1 (AFS score≥5);
2. Scheduled for hysteroscopic adhesiolysis;
3. Agreed to have two follow-up hysteroscopy; and
4. Written, informed consent obtained.

Exclusion Criteria:

1. Received estrogen therapy within 3 months of enrollment;
2. Suffering from leiomyoma, polyps, cancer, or polycystic ovarian syndrome (PCOS);
3. History of genital tuberculosis; and
4. Contraindication for estrogen therapy.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fu Xing Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- 2mg Estradiol Therapy(Low Dose): 2mg oral E2 (Femoston, Abbott Biologicals B.V.) daily for 21 days, followed by 20mg dydrogesterone daily for the last 10 days of hormone treatment.
  Femoston: Femoston is a Complex Packing Estradiol Tablets and Estradiol and Dydrogesterone.
- 6mg Estradiol Therapy(High Dose): 6mg oral E2 (Femoston, Abbott Biologicals B.V.) daily for 21 days, followed by 20mg dydrogesterone daily for the last 10 days of hormone treatment.
  Femoston: Femoston is a Complex Packing Estradiol Tablets and Estradiol and Dydrogesterone.
Period: Overall Study
Arm/Group | 2mg Estradiol Therapy(Low Dose) | 6mg Estradiol Therapy(High Dose)
Started | 70 | 71
Completed | 59 | 62
Not Completed | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- 2mg Estradiol Therapy(Low Dose): mean Age(y):31.9 Gender:Female BMI:21.2 mean Number of miscarriage: 2.3
  BMI=body mass index
- 6mg Estradiol Therapy(High Dose): mean Age(y):32.3 Gender:Female BMI:21.0 mean Number of miscarriage: 2.1
  BMI=body mass index
- Total: Total of all reporting groups
Arm/Group | 2mg Estradiol Therapy(Low Dose) | 6mg Estradiol Therapy(High Dose) | Total
Number analyzed (Participants) | 59 | 62 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (5.0) | 32.3 (4.1) | 32.3 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 62 | 121
  Male | 0 | 0 | 0
Parity [Mean (Standard Deviation); unit: times] — Parity means the number of past deliveries.
  times | 0.2 (0.4) | 0.2 (0.4) | 0.2 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: the AFS Score at Second-look Hysteroscopy
Description: The AFS score is based on the American Fertility Society (AFS) Classification of Intra-uterine adhesions( 1988 version)The total range of AFS score is from 0 to 12, and the higher the score is, the worse the outcome is.
Time Frame: 1 months after the surgery
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | 2mg Estradiol Therapy(Low Dose) | 6mg Estradiol Therapy(High Dose)
Number analyzed (Participants) | 59 | 62
units on a scale | 1.6 (1.4) | 1.9 (1.6)
Statistical Analysis 1: Comparison: 2mg Estradiol Therapy(Low Dose) vs 6mg Estradiol Therapy(High Dose); Test type: Superiority or Other; p > 0.05, t-test, 2 sided

2. Secondary Outcome: the AFS Score at Third-look Hysteroscopy
Description: as for outcome 1
Time Frame: 2 months after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2mg Estradiol Therapy(Low Dose) | 6mg Estradiol Therapy(High Dose)
Number analyzed (Participants) | 59 | 62
units on a scale | 1.0 (1.1) | 1.2 (1.4)

3. Secondary Outcome: Participants With Improvement of Menstrual Pattern at Third-look Hysteroscopy
Description: The menstrual pattern is clarified as four types which includes amenorrhea, scant spotting, light period, normal period. The menstrual pattern of every participant was recored and compared with herself (before and 3 months after surgery). The number showed below is patients whose menstrual pattern had improved after surgery and estrogen therapy.
Time Frame: 3 months after surgery
Measure: Number; unit: participants
Arm/Group | 2mg Estradiol Therapy(Low Dose) | 6mg Estradiol Therapy(High Dose)
Number analyzed (Participants) | 59 | 62
participants | 38 | 44

ADVERSE EVENTS:
Time Frame: 2 months after estradiol therapy
Arm/Group | 2mg Estradiol Therapy(Low Dose) | 6mg Estradiol Therapy(High Dose)
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/62
Other Adverse Events (participants affected / at risk) | 6/59 | 11/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2mg Estradiol Therapy(Low Dose) (N=59) | 6mg Estradiol Therapy(High Dose) (N=62)
nauseated and bloated (Reproductive system and breast disorders) | 6 | 10
abnormal liver function (Hepatobiliary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes